CLINICAL TRIAL: NCT02854358
Title: Efficacy of Traditional Persian Medicine Preparation Versus Artificial Saliva for Radiation Induced Xerostomia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shiraz University of Medical Sciences (Other)
Collaborators: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, seyed hamdollah mosavat, assisstant professor, Shiraz University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CT.9732
Record Dates: First submitted 2016-07-31; First posted 2016-08-03 (Estimated); Last update posted 2016-08-03 (Estimated); Status verified 2016-07

CONDITIONS: Xerostomia; Head and Neck Cancers
MeSH Terms: conditions — Xerostomia; Head and Neck Neoplasms | interventions — Saliva, Artificial

ARMS (2):
- control (Active Comparator): In the control group, patients received Hypozalix (artificial saliva)spray three times per day for a period of four weeks.
  Interventions: Drug: Hypozalix spray (artificial saliva)
- intervention (Experimental): Patients in intervention group received sachets containing 4 grams of mixed powder of A. digitata and M. sylvestris (in a proportion of 1:1), three times per day for a period of four weeks
  Interventions: Drug: mixed powder of A. digitata and M. sylvestris

INTERVENTIONS:
Drug: mixed powder of A. digitata and M. sylvestris
  Other Names: Traditional Persian Medicine preparation
  Arms: intervention
Drug: Hypozalix spray (artificial saliva) — Hypozalix spray (artificial saliva)
  Arms: control

SUMMARY:
Head and neck cancers(HNC) is one of the most common cancers worldwide. Xerostomia is one of the most common side effect of radiation therapy among patients with HNC. Mouth dryness significantly impairs patients' quality of life (QOL).

HNC.Regarding to traditional use of A. digitata and M. sylvestris in addition to known their beneficial effects in recent studies, we decided to design a randomized, controlled clinical trial to try to evaluate efficacy of the these herbs in QOL of HNC patients with radiation induced xerostomia

ELIGIBILITY:
Inclusion Criteria:

* patients with head and neck cancer who had grade 1 and 2 xerostomia (based on the Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0) and finished radiotherapy at least two months before the study(22).

Exclusion Criteria:

* history of connective tissue disorder (e.g., Sjogren) other medical causes of xerostomia (such as diabetes, bowel and renal diseases), using antidepressants drugs, recurrence of cancer, end stage cancer, pregnancy, lactation history of hypersensitivity or allergy to A. digitata and M. sylvestris

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-03; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
changes in patients' quality of life | 4 weeks
  changes in patients' quality of life assessed by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire|(EORTC QLQ-H&N 35)

REFERENCES:
- [Derived] Heydarirad G, Rezaeizadeh H, Choopani R, Mosavat SH, Ameri A. Efficacy of a traditional Persian medicine preparation for radiation-induced xerostomia: a randomized, open-label, active-controlled trial. J Integr Med. 2017 May;15(3):201-208. doi: 10.1016/S2095-4964(17)60333-9. PMID 28494850